CLINICAL TRIAL: NCT05108142
Title: Impact of Resistant Starch Type-3 on Glucose Metabolism and Appetite in Healthy Adult Males
Brief Title: Resistant Starch Type-3, Glucose Metabolism and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Maha Alhussain, Principal Investigator, King Saud University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19/01008
Record Dates: First submitted 2021-10-13; First posted 2021-11-04 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Resistant Starch
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control meal (Experimental): Participants were asked to visit the lab and consume the control meal (hot, freshly cooked pasta)
  Interventions: Other: Dietary intervention
- Resistant starch meal (Experimental): Participants were asked to visit the lab and consume the resistant starch meal (re-heated pasta)
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — fresh, hot pasta and re-heated pasta

SUMMARY:
Resistant starch (RS) is considered to have many of the same health benefits as dietary fiber. The aim of this study was to examine the effects of RS3 on postprandial glycemic and insulinemic responses and appetite.

Healthy males (aged 18-35 years) participated in this study. Subjects were provided meals in the laboratory after overnight fasting on two separate occasions, at least 1 week apart. On each laboratory visit, subjects were given either a control meal (COM) or an RS3 meal (RSM). Both meals during the two visits consisted of vegetarian pasta and were matched for energy intake, composition, ingredients, and amount, but were prepared in different ways. The COM was hot, freshly cooked pasta, while the RSM was re-heated pasta that had been cooked the previous day and chilled overnight. Blood samples and subjective appetite ratings were collected at fasting and for a period of 3 h after meal consumption (i.e., 15-min intervals for glucose and 30-min intervals for insulin, ghrelin, and subjective appetite).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Aged between 18 and 40 years
* Normal weight (BMI 18.5-24.9 kg/m2)
* No history of serious disease or currently taking any medications
* Not dieting or seeking to lose weight.

Exclusion Criteria:

* Smokers
* Allergy to gluten-containing products, lactose intolerance, or dairy allergy
* Particular dislike to any of the foods provided during the study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in fasting and postprandial blood glucose concentrations (n=8) | 3 hours
  Fasting and postprandial blood glucose assessed with the use of a portable monitor (Accu-Chek) during laboratory visits (before and 3 hours following the meal consumption in the two visits).

SECONDARY OUTCOMES:
Changes in of fasting and postprandial serum insulin concentrations (n=8) | 3 hours
  Fasting and postprandial serum insulin assessed using a commercial kit during laboratory visits (before and 3 hours following the meal consumption in the two visits)
Changes in subjective appetite ratings (Visual Analogue Scale) (n=8) | 3 hours
  Subjective appetite ratings were assessed during laboratory visits (before and 3 hours following the meal consumption in the two visits) with the use of paper-based visual analog scales with words anchored at each end of a 100-mm horizontal line that expressed the most-positive rating and the most-negative rating for a question. The questions were in the form of "How (rating) do you feel?" (with ratings of hungry, satisfied, and full), "How much of a desire to eat?" and "How much do you think you can eat?"
Changes in fasting and postprandial plasma ghrelin concentrations (n=8) | 3 hours
  Fasting and postprandial ghrelin assessed using a commercial kit during laboratory visits (before and 3 hours following the meal consumption in the two visits)

CONTACTS AND LOCATIONS:
Locations (1):
- Maha Alhussain, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided